CLINICAL TRIAL: NCT06955390
Title: An Exploratory Clinical Study of HRS-4642 in Combination With SHR-A2102 for the Treatment of Advanced Solid Tumors
Brief Title: Clinical Trial of HRS-4642 Plus SHR-A2102 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-HRS4642-SHRA2102
Record Dates: First submitted 2025-04-20; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR-A2102+HRS-4642
  Interventions: Drug: SHR-A2102+HRS-4642

INTERVENTIONS:
Drug: SHR-A2102+HRS-4642 — A fixed dose was used for SHR-A2102,HRS-4642 can be dose adjusted.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of HRS-4642 combined with SHR-A2102 in the treatment of advanced solid tumors

DETAILED DESCRIPTION:
This study is a prospective, single-arm, exploratory clinical trial. It plans to enroll patients with advanced solid tumors , treating them with HRS-4642 in combination with SHR-A2102. The entire study is divided into two stages: a safety run-in period and an efficacy exploration period.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to give informed consent, have signed informed and able to comply with the treatment plan to visit the tests and other procedural requirements
2. The age of signing the informed consent is from 18 to 75 years old, regardless of gender
3. Subjects with pathologically confirmed locally advanced unresectable or metastatic solid tumors
4. The ECOG score is 0 or 1
5. Expected survival ≥12 weeks
6. At least one measurable lesion according to RECIST v1.1 criteria
7. Good level of organ function
8. Male subjects whose partners are women of childbearing age and female subjects who are fertile are required to use highly effective contraceptive methods

Exclusion Criteria:

1. subjects with uncontrolled or active brain metastasis；
2. subjects with clinical significant lung disease;
3. subjects with history of autoimmune diseases;
4. Known active hepatitis B or C infection;
5. Subjects with severe cardiovascular and cerebrovascular diseases
6. Uncontrolled tumor-related pain
7. Severe infections that require intravenous antibiotic, antiviral or antifungal control
8. Clinically symptomatic moderate to severe ascites; Uncontrollable or moderate or above pleural effusion, pericardial effusion
9. Received anti-tumor therapy 4 weeks prior to initiation of study treatment.
10. Known allergic to any compound of SHR-A2102 or HRS-4642
11. Other serious accompanying illnesses, which, in the investigator's assessment, could seriously adversely affect the safety of the treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity(DLT) | At the end of Cycle 1 (each cycle is 14 days)
  one or more unacceptable toxic reactions that occur after administration, leading to an inability to further increase the dose or extend the dosing cycle.
Objective Response Rate (ORR) | up to 1 year
  the proportion of patients with a confirmed complete response or partial response on two consecutive occasions≥4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  the time from treatment initiation to the first disease progression or death from any cause
Overall survival(OS) | up to 2 year
  the time from treatment initiation until death from any reason
Disease Control Rate (DCR) | up to 1 year
  the proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD)
Duration of response (DoR) | up to 1 year
  Assessed by Investigator According to RECIST v1.1
Incidence and severity of adverse events (AE) and serious adverse events (SAE) and laboratory | Begin from sign the ICF until the end of the safety follow-up period，Up to approximately 2 years.
  Assess safety and tolerability by way of adverse events (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Professor, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No